CLINICAL TRIAL: NCT04190979
Title: Clinical Application of the Medyria TrackCath System in Endovascular Repair of Abdominal Aortic Aneurysms (AAA) - A Prospective Multi-centre Clinical Trial.
Brief Title: Clinical Application of the Medyria TrackCath System in Endovascular Repair of Abdominal Aortic Aneurysms (AAA)
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medyria AG (Industry)
Collaborators: StatConsult Gesellschaft für klinische und Versorgungsforschung mbH (Unknown); Axxos GmbH (Unknown); Worldwide Clinical Trials (Other); Medical Mind RCS GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-000 214
Record Dates: First submitted 2019-11-14; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracoabdominal; Acute Renal Failure; Acute Kidney Injury; Acute Kidney Failure; Acute Renal Insufficiency
Keywords: Endovascular aneurysm repair; EVAR; AAA; Cannulation; Blood Flow Velocity
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracoabdominal; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): TrackCath
  Interventions: Device: Medyria TrackCath System

INTERVENTIONS:
Device: Medyria TrackCath System — The TrackCath System is a non-implantable device and consists of the TrackCath Catheter and the TrackCath Equipment. It is designed to support the successful positioning of third-party guidewires and catheters in the arterial vasculature to detect and cannulate side branches during endovascular aneurysm repair procedures through the measurement of real-time blood flow velocity changes.

SUMMARY:
Pre-market, single-arm, prospective, open-label, multi-center clinical trial aimed at assessing the safety and the performance of the Medyria TrackCath system in patients undergoing endovascular intervention.

DETAILED DESCRIPTION:
Pre-market, single-arm, prospective, open-label, multi-center clinical trial aimed at assessing the safety and the performance of the Medyria TrackCath system in patients above the age of 18 years who have been diagnosed with aneurysms in the thoracoabdominal (TAAA) or abdominal (AAA) aorta and require endovascular intervention.

The TrackCath System is a non-implantable disposable device, intended to measure real-time changes in the Blood Flow Velocity and to provide a pathway for delivering third-party guidewires and/or catheters.

Following patient consent, data is collected until discharge.

To reach 80% power, a total number of 32 patients (minimum 42 target orifices) is scheduled, including a minimum of 8 roll-in patients for the training phase, which comprises at least two successful cases per center.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and understood the approved Informed Consent form and is able to meet the proposed study proceedings (CIP).
* Patient is ≥18 years of age
* Need for standard or complex EVAR of AAA according to the relevant guidelines:
* Asymptomatic aneurysms with a diameter > 55mm in men and > 50 mm in woman
* Aneurysm-growth exceeds 10mm/year
* Patient requires at least one cannulation during which requires at least one cannulation (e.g. fenestration of endograft, side-branch and/or contralateral leg of endograft)

Exclusion Criteria:

* Patient is generally contraindicated for EVAR
* Patient requires an emergency surgery
* Patient with an increased risk of aneurysm rupture or saccular aneurysm, aneurysm with isolated wall protuberances or penetrating aortic ulcer
* Patient with a dissecting acutely ruptured or leaking aneurysm or an acute vascular injury caused by a trauma
* Patient with stroke or transient ischemic attack (TIA) within the last 6 months prior to baseline
* Patient with myocardial infarction (MI) with the last 3 months prior to baseline
* Patient with acute or chronic renal failure (including dialysis); Creatinine > 2.00 mg/dl or > 182 µmol/L
* Patient with co-morbidities that constitutes an unacceptable risk (for example chronic obstructive pulmonary disease (COPD), liver failure, immunosuppression, polyneuropathy and hematological diseases)
* Patient with bleeding history or coagulopathy
* Patient with contraindication or allergies to take anticoagulants, antiplatelet drugs or contrast media
* Life expectancy of less than 5 years
* Female patient that is pregnant, is planning on becoming pregnant in the next month or is breastfeeding
* Patient with inability to obtain vascular access
* Patient has an active local or systemic infection
* Patient is currently participating in another investigational study where the endpoints have not yet been achieved
* Patient has a mental illness, and/or been diagnosed as clinically depressed or belongs to a vulnerable population (e.g., prisoner, severe drug abuser, developmentally disabled) that would compromise the ability to provide informed consent.
* Patient has an obstructed or inadequate vasculature by means of tortuous anatomy hindering the TC catheter to reach target orifice(s)
* Patient has an elevated risk of plaque dislodgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-17 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Procedural Success Rate | Intra-operative
  Successful TrackCath delivery of the distal end of the guidewire or of the 4 French catheter to the selected targeted orifice(s).
Primary Safety (All SADEs) | Up to discharge (expected to be within 1 month)
  Occurrence of Serious Adverse Device Effects (SADE)

SECONDARY OUTCOMES:
Secondary Safety (All AEs) | Up to discharge (expected to be within 1 month)
  All Adverse Events
Procedural Parameters (contrast dye) | Intra-operative
  Amount of contrast dye used (ml)
Procedural Parameters (procedural times) | Intra-operative
  Exposure time to X-ray (min); total duration of the procedure (min); duration of the target orifice identification and cannulation (min).
Procedural Parameters (Blood flow velocity) | Intra-operative
  Blood flow velocity changes between above orifice and at orifice (m/s).
Surgeon satisfaction rate | Intra-operative
  Surgeon satisfaction on the use of the TrackCath catheter and the Blood Flow Velocity sensor, expressed on a scale from 1 (very bad) to 5 (very good).

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Schelzig, Prof. Dr., Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (4):
- Germany (4):
  - Universitätsklinikum RWTH Aachen, Aachen
  - Heinrich-Heine University Düsseldorf, Düsseldorf
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Universitätklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No